CLINICAL TRIAL: NCT06940440
Title: IFx-Hu2.0 As An Adjunctive Therapy To Pembrolizumab In Checkpoint Inhibitor Naïve Subjects With Advanced Or Metastatic Merkel Cell Carcinoma
Brief Title: IFx-Hu2.0 As An Adjunctive Therapy To Pembrolizumab In Advanced Or Metastatic Merkel Cell Carcinoma (MCC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TuHURA Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC 2023-01
Expanded Access: NCT04853602 (Available)
Record Dates: First submitted 2025-04-03; First posted 2025-04-23 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Advanced Or Metastatic Merkel Cell Carcinoma
Keywords: Metastatic; Advanced; Merkel Cell Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Merkel Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IFx-Hu2.0 (Experimental): Subjects will receive IFx-Hu2.0 (0.1 mg) as a visceral lesion injection in a single lesion once per week for three consecutive weeks. KEYTRUDA® (pembrolizumab) (200 mg) will be administered intravenously (IV) on Visit 1 (within 48 hours from the first IFx-Hu2.0 injection) then every three weeks for approximately six months, until disease progression or unacceptable immune related toxicity.
  Interventions: Drug: IFx-Hu2.0; Drug: Pembrolizumab

INTERVENTIONS:
Drug: IFx-Hu2.0 — Therapeutic Classification:
  • Innate immune agonist
  Route of Administration:
  • Intralesional
  Other Names: pAc/emm55
Drug: Pembrolizumab — Therapeutic Classification:
  • Immunotherapy (Immune checkpointinhibitor)
  Route of administration:
  • Intravenous (IV) infusion
  Other Names: KEYTRUDA

SUMMARY:
This Phase 1, multicenter, open-label trial will assess the safety and feasibility of IFx-Hu2.0 as adjunctive therapy to pembrolizumab in adult patients (≥18 years) with non-cutaneous Merkel Cell Carcinoma. Nine subjects will receive IFx-Hu2.0 as a visceral lesion injection in a single lesion followed by pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Life expectancy equal to or greater than six months.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status < 2.
4. Active disease measurable by CT or MRI, measurable lesions are lesions that can be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded).
5. Must be recurrent and/or unresectable Stage III or Stage IV American Joint Committee on Cancer (AJCC) (8th edition) and have histologically confirmed Merkel cell carcinoma

   a. Must have at least one visceral injectable lesion equal to or greater than 3 mm
6. Subject should be CPI naïve i.e., no prior therapy with CPI including but not limited to Pembrolizumab, avelumab, ipilimumab, nivolumab.
7. Tumor tissue from an archival core biopsy or resected site of disease must be provided for biomarker analyses. If archival tissue is not available, then a new biopsy should be performed.
8. Adequate hematological, hepatic, and renal function according to laboratory ranges and medical criteria defined within the study protocol.

Exclusion Criteria

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with protocol requirements.
2. Subjects with active brain metastases, with the exception of treated brain metastases that have imaging proving stability at least 4 weeks after treatment, no new metastases, and not requiring steroids.
3. Subjects with recurrent resectable MCC
4. Subjects who have received prior systemic chemotherapy
5. Pregnant or breastfeeding females and females desiring to become pregnant or breastfeed within the timeframe of this study.
6. Active, known, or suspected autoimmune disease. Potential subjects with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. Low grade autoimmune toxicity is NOT an exclusion under this criterion.
7. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of IFx-Hu2.0 administration. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety | 28 days from last dose of IFx-Hu2.0
  Safety is defined as the absence of any grade 3-5, treatment-related Adverse Events (AEs) per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 from first injection Day 1 to 28-day follow-up after the final dose of IFx-Hu2.0.
Feasibility | 28 days from last dose of IFx-Hu2.0
  Feasibility is defined as the ability to treat ≥50% of subjects (i.e. 5/9) in the per-protocol analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Brohl, MD, Principal Investigator — Collaborator
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin